CLINICAL TRIAL: NCT02135627
Title: TC-325 (HEMOSPRAY™) VS. CURRENT STANDARD OF CARE IN MANAGING MALIGNANT GASTROINTESTINAL BLEEDING: A PILOT STUDY TO INFORM A RANDOMIZED CONTROLLED TRIAL.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: ASGE (Unknown)
Responsible Party: Principal Investigator, Alan Barkun, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-251-BMD
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: MALIGNANT GASTROINTESTINAL BLEEDING
MeSH Terms: interventions — Epinephrine; Sclerotherapy; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Experimental): Current standard endoscopic therapy such as epinephrine injection, sclerotherapy, mechanical (endoclip). contact electrocautery/thermal, and non-contact electrocalcautery (APC) ± radiation therapy, angioembolization, and/or surgery.
  Interventions: Other: Current standard therapy
- TC-325 (Active Comparator): TC-325 monotherapy on initial endoscopy ± radiation therapy, angioembolization, and/or surgery.
  Interventions: Drug: TC-325 monotherapy on initial endoscopy ± radiation therapy, angioembolization, and/or surgery.

INTERVENTIONS:
Drug: TC-325 monotherapy on initial endoscopy ± radiation therapy, angioembolization, and/or surgery.
  Arms: TC-325
Other: Current standard therapy
  Other Names: epinephrine injection,; sclerotherapy,; mechanical (endoclip).; contact electrocautery/thermal; non-contact electrocalcautery (APC) ± radiation therapy,; angioembolization,; surgery
  Arms: Control group

SUMMARY:
Introduction: Gastrointestinal (GI) bleeding arising from malignant tumors is increasingly recognized as a result of oncological advances and improved detection methods, and stems from local vessel damage and tumor invasion with associated derangements in the hemostatic system(1, 2). Although conventional endoscopic hemostasis methods improve outcomes in UGIB due to peptic ulcers and other non-variceal benign bleeding lesions of the upper, and perhaps the lower GI tract, data on their use in hemorrhagic, upper or lower gastrointestinal neoplasms are scarce and associated with varying success in initial hemostasis and high rebleeding rates(3-7). Other recognized single or multimodality treatment approaches include radiation therapy, interventional angiography, and surgery. All exhibit disappointing rebleeding rates, and in the case of emergency surgery, high mortality(4, 8-11). Challenges associated with bleeding tumors include hematological derangements such as thrombocytopenia, disseminated intravascular coagulation, and neutropenia, as well as the endoscopic manipulation of friable, diffusely bleeding surfaces when attempting hemostasis(2, 12, 13). The recent advent of TC-325 (HemosprayTM) to Canada, Europe and Asia - referred henceforth as TC-325 - may provide a highly adapted novel endoscopic hemostatic therapeutic alternative for this refractory clinical entity, with promising uncontrolled observations having just been published by our group(13) and others(14). More robust controlled evaluative data are now needed. We propose to study the use of TC-325 in upper and lower malignant GI bleeding compared to contemporary standard of care, and more specifically seeks funding for a pilot study to inform a subsequent peer-review application for a larger, more definitive randomized clinical trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* able to comprehend the trial and provide written informed consent in French or English, or a close relative with power of attorney
* Patients who present with an upper or lower GI bleeding with a known luminal GI malignancy diagnosed within the past two years will be considered for enrolment. Endoscopic confirmation of an active GI bleed arising from a malignant tumor will be required for final inclusion
* Rebleeding in patients who presented with acute GIB with initial endoscopy suggesting a malignant source based on endoscopic appearance who have not been treated previously with TC-325 will also be included

Exclusion Criteria:

* Refused by patient
* Pregnancy
* Bleeding from non-malignant GI sources such as gastritis/duodenitis, Mallory Weiss syndrome, peptic ulcer disease, varices, vascular malformations, radiation proctitis, polyps, hemorrhoids, and diverticulosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Hemostasis | 3 minutes after endoscopic therapy
  The main outcome will be rate of immediate hemostasis with application of TC-325 or conventional hemostatic therapy. Immediate hemostasis is defined as the absence of bleeding following 3 minutes of observation after endoscopic therapy.

SECONDARY OUTCOMES:
Rebleeding | 1, 3, 30, 90 and 180 days following randomization
  Rebleeding following randomization
Transfusion | 30 days after randomization
  transfusion requirements
length of ICU admission | 180 days
  need for admission to and length of stay in a monitored care unit
Length of hospitalization | 180 days
  Total length of hospitalization
Complications | day 1
  Complications associated with endoscopy
Additional treatment modalities | 30 days
  Rates of use of additional treatment modalities to stop persistent bleeding or rebleeding after the index event
Mortality | 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Chen YI, Wyse J, Lu Y, Martel M, Barkun AN. TC-325 hemostatic powder versus current standard of care in managing malignant GI bleeding: a pilot randomized clinical trial. Gastrointest Endosc. 2020 Feb;91(2):321-328.e1. doi: 10.1016/j.gie.2019.08.005. Epub 2019 Aug 19. PMID 31437456